CLINICAL TRIAL: NCT02752152
Title: A Randomized Study to Compare Three Counseling Strategies and Evaluate the Efficacy of Reminders for Regular HIV, Hepatitis B and C, and Syphilis Testing
Brief Title: Counseling and Reminders for Regular HIV and STIs Screening
Acronym: Napneung-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recherche pour le Developpement (Other Government)
Collaborators: Chiang Mai University (Other); Expertise France (Other)
Responsible Party: Principal Investigator, GONZAGUE JOURDAIN, PHPT research Team, Institut de Recherche pour le Developpement
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Napneung-1
Record Dates: First submitted 2016-04-22; First posted 2016-04-26 (Estimated); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: HIV, Hepatitis B, Hepatitis C and Syphilis Infections
Keywords: Counseling; Reminder; Early diagnosis
MeSH Terms: conditions — Hepatitis B; Hepatitis C; Disease | interventions — Appointments and Schedules

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Computer-assisted counseling (Experimental): Computer-assisted informational/educational interactive session followed by an interactive face-to-face session to discuss personal issues with a counselor as needed
  Interventions: Behavioral: Computer-assisted counseling; Behavioral: Appointment + reminder; Behavioral: Reminder; Behavioral: No appointment and no reminder
- On-demand counseling (Experimental): The counselor asks whether the participant has any questions
  Interventions: Behavioral: On-demand counseling; Behavioral: Appointment + reminder; Behavioral: Reminder; Behavioral: No appointment and no reminder
- Standard counseling (Active Comparator): Interactive face-to-face counseling session
  Interventions: Behavioral: Standard counseling; Behavioral: Appointment + reminder; Behavioral: Reminder; Behavioral: No appointment and no reminder
- Appointment + reminder (Experimental): Make appointment and send SMS reminder
  Interventions: Behavioral: Computer-assisted counseling; Behavioral: On-demand counseling; Behavioral: Standard counseling; Behavioral: Appointment + reminder
- Reminder only (Experimental): Send SMS reminder only
  Interventions: Behavioral: Computer-assisted counseling; Behavioral: On-demand counseling; Behavioral: Standard counseling; Behavioral: Reminder
- No appointment and no reminder (Active Comparator): No appointment and no SMS reminder sent
  Interventions: Behavioral: Computer-assisted counseling; Behavioral: On-demand counseling; Behavioral: Standard counseling; Behavioral: No appointment and no reminder

INTERVENTIONS:
Behavioral: Computer-assisted counseling — The counselor opens the computer-assisted information/educational interactive counseling program on the tablet computer and invites the participant to use the program.
  Arms: Appointment + reminder; Computer-assisted counseling; No appointment and no reminder; Reminder only
Behavioral: On-demand counseling — The counselor only invites the participants to ask questions about HIV and other STIs.
  Arms: Appointment + reminder; No appointment and no reminder; On-demand counseling; Reminder only
Behavioral: Standard counseling — The counselor gives face-to-face general information/education
  Arms: Appointment + reminder; No appointment and no reminder; Reminder only; Standard counseling
Behavioral: Appointment + reminder — Has an appointment and receive reminders for further testing
  Arms: Appointment + reminder; Computer-assisted counseling; On-demand counseling; Standard counseling
Behavioral: Reminder — Only receive reminders for further testing
  Arms: Computer-assisted counseling; On-demand counseling; Reminder only; Standard counseling
Behavioral: No appointment and no reminder — No appointment and no reminders for further testing
  Arms: Computer-assisted counseling; No appointment and no reminder; On-demand counseling; Standard counseling

SUMMARY:
Counseling intervention:

Primary objective: to evaluate and compare, in at-risk populations, the efficacy of three different counseling methods in terms of propensity to come back for a HIV re-test. Secondary objectives: to evaluate and compare the efficacy of the counseling methods in terms of reported risk behavior and HIV knowledge as well as their acceptability and cost-effectiveness; describe the distribution of duration from HIV primary infection to detection; and estimate the prevalence of chronic hepatitis B and C, and syphilis in HIV-uninfected participants of targeted populations.

Reminder intervention Primary objective: to evaluate and compare, in at-risk individuals who require frequent testing, the efficacy of reminders in terms of propensity to come back for a HIV re-test within 7 months.

Secondary objective: to assess the cost-effectiveness of reminders.

The interim analyses have shown that that some strategies are better than the others and the Advisory Committee recommended to use only the most efficient strategies (Computer assisted counseling and Scheduling an appointment and sending reminder to clients).

In addition, CD4 cell count normal ranges in 30 HIV uninfected individuals in Thailand will be assessed. Transient elastometry (FibroScan) will be used to assess liver fibrosis in participants with and without viral hepatitis.

DETAILED DESCRIPTION:
The study will be presented to clients, who will be asked to formally consent to participate. Clients residing or working in Thailand and able to communicate with the counselor will be eligible. Foreigners staying in Thailand for vacation or retirement will be excluded, except if presenting together with their partner who is otherwise eligible for the study. At each visit, participants will be proposed an appointment for a re-test. If they wish, the study team will send them reminders.

At the first visit, participants will be randomly assigned to one of three different methods for counseling on HIV, hepatitis B and C, and syphilis: standard face-to-face counseling, computer-assisted informational/educational counseling, or on-demand counseling (the counselor invites the participant to ask questions). Participants will then be randomly assigned to one of three reminder strategies: Appointment+reminder, Reminder only, or No appointment and no reminder.

At each visit, blood sample will be collected to test for HIV, hepatitis B and C, and syphilis. Laboratory examinations will be free of charge for all participants. After the blood draw, participants will be invited to complete a questionnaire to assess their knowledge, attitudes and practices with regard to HIV and other infections. Test results will then be provided. In case of confirmed HIV infection, participants will be provided with further counseling, CD4 cell count measurement and referral options for immediate treatment. Blood samples collected during the study for the diagnosis will be stored for determination of the Fiebig stage (duration since HIV primary infection), evaluation of transmitted HIV drug resistance (sequencing) and investigation of viral transmission networks.

In a substudy, we will compare liver fibrosis assessed by transient elastometry and serum biomarkers (i.e. APRI and FIB-4) in Napneung participants with HBsAg and those with anti-HCV antibodies, and compare the measures with that obtained in participants negative for these tests.

The interim analyses have shown that that some strategies are better than the others and the Advisory Committee recommended to use only the most efficient strategies (Computer assisted counseling and Scheduling an appointment and sending reminder to clients). Thus the accrual to the arms "No appointment, no reminder" and "Reminder only" has been discontinued on 12 January 2019.

Following the published of CD4 cell count normal ranges in HIV uninfected individuals in Thailand since 1997 (Vithayasai, Sirisanthana, Sakonwasun, & Suvanpiyasiri, 1997), It is unknown whether these norms have changed in relation to changes in nutritional status and lifestyle in young adults. We will assess the number of CD4 cells/mL in the blood of the first 30 HIV-uninfected female and the first 30 HIV-uninfected male clients aged less than 26 years to determine whether there is a trend for an increase in young people due to the changes in nutrition and lifestyle during the last decades. This sub-study will be conducted from 1 February 2019 to 31 January 2021.

ELIGIBILITY:
Inclusion Criteria:

* Residing or working in Thailand
* Able to communicate with the counselor
* Adults (>= 18 years old)

Exclusion Criteria:

* Foreigners staying in Thailand for vacation or retirement, except if they are presenting together with their partner staying permanently in Thailand or working in Thailand
* Couples requesting a couple counseling session
* HIV-positive participants (based on the client declaration)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1961 (Actual)
Dates: Start 2015-12-09 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2020-10-18 (Actual)

PRIMARY OUTCOMES:
Percentage of participants from at-risk populations coming for a HIV re-test | Within 7 months following the first visit
  Number of participants having a re-test divided by number of at-risk participants

CONTACTS AND LOCATIONS:
Overall Officials: Gonzague Jourdain, MD. PhD, Principal Investigator — IRD
Locations (3):
- Thailand (3):
  - Faculty of Associated Medical Sciences, Chiang Mai University, Chiang Mai
  - MAP Foundation testing facility, Chiang Mai
  - Special clinic of Chiangrai Prachanukroh Hospital, Chiang Rai

IPD SHARING:
Plan to Share IPD: Undecided
To be discussed with the steering committee

REFERENCES:
- [Derived] Salvadori N, Decker L, Ngo-Giang-Huong N, Mary JY, Chevret S, Arunothong S, Adam P, Khamduang W, Samleerat T, Luangsook P, Suksa-Ardphasu V, Achalapong J, Rouzioux C, Sirirungsi W, Jourdain G. Impact of Counseling Methods on HIV Retesting Uptake in At-Risk Individuals: A Randomized Controlled Study. AIDS Behav. 2020 May;24(5):1505-1516. doi: 10.1007/s10461-019-02695-2. PMID 31605294
- See also: Official study site for the recruitment — https://www.napneung.org/
- See also: Official facebook page for the recruitment — https://th-th.facebook.com/napneung